CLINICAL TRIAL: NCT01708889
Title: An Open-label, Single Dose Study to Evaluate the Pharmacokinetics, Safety, and Tolerability of BMS-914143 in Subject With Normal Renal Function and Subjects With Mild, Moderate, Severe, and End-stage Renal Dysfunction
Brief Title: Pharmacokinetic Study of BMS-914143 in Participants With Normal Renal Function and Mild, Moderate, Severe and End-stage Renal Dysfunction
Acronym: PK
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None
Other Study IDs: AI452-019
Record Dates: First submitted 2012-10-16; First posted 2012-10-17 (Estimated); Last update posted 2013-06-05 (Estimated); Status verified 2013-06

CONDITIONS: Chronic Hepatitis B Virus Infection; Chronic Hepatitis C Virus Infection
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — peginterferon lambda-1a

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- Group 1: BMS-914143 (eGFR ≥ 80 mL/min/1.73 m2) (Experimental): BMS-914143 (Peginterferon Lambda-1a) single 180 µg Solution, Subcutaneous injection for subjects with normal renal function with eGFR ≥ 80 mL/min/1.73 m2
  Interventions: Biological: BMS-914143 (Peginterferon Lambda-1a)
- Group 2: BMS-914143 (eGFR 60 to 79 mL/min/1.73 m2) (Experimental): BMS-914143 (Peginterferon Lambda-1a) single 180 µg Solution, Subcutaneous injection for subjects with mild renal dysfunction with eGFR 60 to 79 mL/min/1.73 m2
  Interventions: Biological: BMS-914143 (Peginterferon Lambda-1a)
- Group 3: BMS-914143 (eGFR 30 to 59 mL/min/1.73 m2) (Experimental): BMS-914143 (Peginterferon Lambda-1a) single 180 µg Solution, Subcutaneous injection for subjects with moderate renal dysfunction with eGFR 30 to 59 mL/min/1.73 m2
  Interventions: Biological: BMS-914143 (Peginterferon Lambda-1a)
- Group 4: BMS-914143 (eGFR 15 to 29 mL/min/1.73 m2) (Experimental): BMS-914143 (Peginterferon Lambda-1a) single 180 µg Solution, Subcutaneous injection for subjects with severe renal dysfunction with eGFR 15 to 29 mL/min/1.73 m2
  Interventions: Biological: BMS-914143 (Peginterferon Lambda-1a)
- Group 5: BMS-914143 (eGFR < 15 mL/min/1.73 m2) (Experimental): BMS-914143 (Peginterferon Lambda-1a) single 180 µg Solution, Subcutaneous injection for subjects with end-stage renal dysfunction with eGFR < 15 mL/min/1.73 m2 (on hemodialysis [HD] or non-HD)
  Interventions: Biological: BMS-914143 (Peginterferon Lambda-1a)

INTERVENTIONS:
Biological: BMS-914143 (Peginterferon Lambda-1a)
  Other Names: Lambda

SUMMARY:
The purpose of this study is to determine the effect of renal impairment on pharmacokinetics (PK) of BMS-914143.

DETAILED DESCRIPTION:
Primary purpose: Protocol designed to evaluate the effect of renal impairment on pharmacokinetics of BMS-914143

ELIGIBILITY:
Inclusion Criteria:

* Normal renal function or mild, moderate, severe or end-stage renal dysfunction

Exclusion Criteria:

* History of uncontrolled or unstable cardiovascular, respiratory, gastrointestinal, hepatic, endocrine, hematopoietic, psychiatric or neurological conditions within 6 months of Lambda administration
* History of chronic liver disease including cirrhosis, hepatitis B virus (HBV), hepatitis C virus (HCV), primary biliary cirrhosis, etc
* History of central nervous system or neuro-psychiatric disease. Subjects with severe depression and/or other uncontrolled psychiatric conditions should not be enrolled in this study
* History of of suicide attempt within the 5 years preceding BMS-914143 administration
* Inability to tolerate subcutaneous injections
* Donation of >400 mL of blood within 8 weeks or plasma within 4 weeks of planned dosing

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2012-09; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Area under the serum concentration-time curve from time 0 extrapolated to infinity [AUC(INF)] of a single 180-μg subcutaneous (SC) dose of Lambda in subjects with normal renal function and subjects with renal dysfunction | 18 time points up to Day 29
Area under the serum concentration-time curve from time 0 to the time of last quantifiable concentration [AUC(0-T)] of a single 180-μg subcutaneous (SC) dose of Lambda in subjects with normal renal function and subjects with renal dysfunction | 18 time points up to Day 29
Maximum observed serum concentration (Cmax) of a single 180-μg subcutaneous (SC) dose of Lambda in subjects with normal renal function and subjects with renal dysfunction | 18 time points up to Day 29
Apparent volume of distribution (Vz/F) of a single 180-μg subcutaneous (SC) dose of Lambda in subjects with normal renal function and subjects with renal dysfunction | 18 time points up to Day 29
Total body clearance (CLT/F) of a single 180-μg subcutaneous (SC) dose of Lambda in subjects with normal renal function and subjects with renal dysfunction | 18 time points up to Day 29

SECONDARY OUTCOMES:
Time to maximum observed serum concentration (Tmax) using serum levels of Lambda | 18 time points up to Day 29
Half life (T-HALF) using serum levels of Lambda | 18 time points up to Day 29
Immunogenicity assessed by serum levels of anti-Lambda antibodies | 5 time points up to Day 43
Safety assessed by Vital signs measurements, electrocardiograms (ECGs), clinical laboratory tests, marked laboratory abnormalities, physical measurements, and adverse events (AEs) | Up to Day 43
Serious adverse events (SAEs) Safety assessed by Vital signs measurements, electrocardiograms (ECGs), clinical laboratory tests, marked laboratory abnormalities, physical measurements, and adverse events (AEs) | Approximately up to Day 73

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (3):
- United States (3):
  - Clinical Pharmacology Of Miami Inc., Miami, Florida
  - Orlando Clinical Research Center, Orlando, Florida
  - New Orleans Center For Clinical Research - Knoxville, Knoxville, Tennessee

REFERENCES:
- See also: BMS clinical trial educational resource — http://www.bms.com/studyconnect/Pages/home.aspx
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx